CLINICAL TRIAL: NCT05802862
Title: A Multi-center, Randomized, Open, Phase III Study of Insulin Degludec/Insulin Aspart Biosimilar (22011) Compared Efficacy and Safety With Insulin Degludec/Insulin Aspart(Ryzodeg) in Chinese Subjects With Type 2 Diabetes
Brief Title: A Study of Insulin Degludec/Insulin Aspart Biosimilar (22011) Compared With Insulin Degludec/Insulin Aspart(Ryzodeg) in Participants With Type 2 Diabetes in China
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22011-DM-301
Record Dates: First submitted 2023-03-06; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 22011 (Experimental)
  Interventions: Drug: Insulin Degludec and Insulin Aspart
- Ryzodeg (Active Comparator)
  Interventions: Drug: Insulin Degludec and Insulin Aspart

INTERVENTIONS:
Drug: Insulin Degludec and Insulin Aspart — administered subcutaneously, once a day

SUMMARY:
The purpose of this study is to see if Insulin Degludec/Insulin Aspart (22011) compared to Insulin Degludec/Insulin Aspart (Ryzodeg) is similar in safety and effect in participants with type 2 diabetes (T2D).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities.
* Male or female, age at least 18 year-old and no more than 75 year-old at the time of signing informed consent.
* Type 2 diabetes mellitus (T2D).
* Body mass index (BMI) higher than 18.0, but below or equal to 35.0 kg/m^2.
* Current treatment for at least 3 months prior to screening with basal insulin/premixed insulin once a day or twice a day with/without oral anti-diabetic drugs (OADs): metformin, alpha-glucosidase inhibitors, dimethylphenylpenicillin dipeptidyl peptidase 4 (DPP-4) inhibitors, sodium-dependent glucose transporter 2 (SGLT-2) inhibitors . For above or equal to 3 months prior to screening subjects should be on a stable dose.
* HbA1c from 7-11.0% both inclusive at screening confirmed by central laboratory analysis.

Exclusion Criteria:

* Have a diagnosis of type 1 diabetes (T1D), or specific type of diabetes other than T2D, for example, injured pancreas, diseases of acromegaly-induced diabetes.
* Have a history of ketoacidosis or hyperosmolar state or coma requiring hospitalization within 6 months prior to screening.
* Have had severe hypoglycemia episodes within 6 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Hemoglobin A1c (HbA1c) | Baseline to Week 24
  HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time

SECONDARY OUTCOMES:
Change From Baseline in Hemoglobin A1c (HbA1c) in Week 12 | Baseline to Week12
  HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time
Percentage of Participant Who Achieved HbA1c<7% and ≤6.5% | Baseline to Week24
  the ratio of participant Who Achieved HbA1c<7% and ≤6.5%
Percentage of Participant Who Achieved HbA1c<7% and ≤6.5% without Hypoglycaemic Episodes | Baseline to Week24
  The ratio of participant Who Achieved HbA1c<7% and ≤6.5% without Hypoglycaemic Episodes
Change From Baseline in Fasting Plasma Glucose(FPG) | Baseline to Week12
  the plasma glucose concentration on an empty stomach
Change From Baseline in Fasting Plasma Glucose(FPG) in Week24 | Baseline to Week24
  the plasma glucose concentration on an empty stomach
Change From Baseline in 7-Point Self-Monitoring Blood Glucose (SMBG) Values | Baseline to Week12
  SMBG 7-point profiles were measured at fasting, 2-hour post morning meal, pre midday meal, 2-hour post midday meal, pre evening meal, 2-hours post evening meal, and bedtime.
Change From Baseline in 7-Point Self-Monitoring Blood Glucose (SMBG) Values in Week24 | Baseline to Week24
  SMBG 7-point profiles were measured at fasting, 2-hour post morning meal, pre midday meal, 2-hour post midday meal, pre evening meal, 2-hours post evening meal, and bedtime.
Change From Baseline in Body weight | Baseline to Week24
  Change in body weight
Number of Treatment-emergent Adverse Events (TEAE) and Serious Adverse Events(SAE) | from baseline to Week25
  Safety

IPD SHARING:
Plan to Share IPD: No